CLINICAL TRIAL: NCT00360204
Title: Improving Health Outcomes for New Mothers and Babies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences Chief, Division of Academic General Pediatrics Vice Chair of Clinical Affairs, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22163; R40 MC 06630-01
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Hyperbilirubinemia; Jaundice; Dehydration; Postpartum Depression
Keywords: Infant health; parenting competence; Home nurse visit; maternal post-partum care; postpartum health utilization; Breastfeeding
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice; Dehydration; Depression, Postpartum; Breast Feeding

INTERVENTIONS:
Behavioral: Home Nurse Visit — Home nurse visit by maternal child health nurse within first 24-48 after post-partum hospital discharge.

SUMMARY:
Because adherence to postnatal care guidelines across the United States (U.S.) is poor, newborns and mothers often are placed at undue risk for adverse medical and social outcomes. This study aims to evaluate an alternative model of care and improve healthcare delivery to and reduce health disparities for "well" newborns and mothers after hospital discharge by using single postnatal home nurse visits. The principal investigator has previously shown a reduction in poor outcomes for infants who receive a home visit after discharge when studied retrospectively. The proposed research will build on the previous study and prospectively evaluate the impact of a single home nursing visit on morbidities and health disparities for newborns and mothers in a randomized, controlled trial involving 1154 mother/infant breastfeeding dyads. Home visits should guarantee detailed assessment during an at-risk period of infancy and motherhood, where medical and social problems can be recognized, anticipated, and/or treated, and can bridge the gap between hospital care and primary care. The investigators' program, The Nurses for Infants Through Teaching and Assessment after the NurserY (NITTANY) Initiative, also will consider the cost-effectiveness of home visitation compared with guidelines-adherent outpatient clinic care.

DETAILED DESCRIPTION:
In the NITTANY Initiative the effectiveness of a single postnatal/postpartum home nurse visit will be evaluated prospectively and compared with outpatient clinic-based care using a randomized, controlled study design. We will attempt to reduce morbidity in the neonatal/postpartum period using a well-timed home visit measured first by a reduction in the need for additional hospital services (inpatient hospitalization and ED visitation) in the first 14 days after delivery. While healthcare utilization may not be the most important health outcome for newborns and mothers from a long-term perspective, the demographic groups at-risk for these outcomes tend to parallel those at greater long-term risk. Also, in the short-term these outcomes may be the most costly ones for insurance providers and can be used in a cost-effectiveness analysis to justify home nurse visits. Readmissions and use of urgent care also may be the most noticeable outcome for clinicians, which should help to modify practice patterns and improve compliance with guidelines for healthcare delivery.

Over a 3-year period we will prospectively enroll a cohort of 1154 "well" singleton newborns and their mothers admitted to the hospital nursery that are most at-risk for readmission based on demographic features. Previous data have indicated those at greatest risk for adverse health outcomes are infants born to breastfeeding mothers and those with less parenting experience. Minorities and Medicaid recipients are more likely to suffer from healthcare disparities. For mothers, morbidities may occur in all socioeconomic groups, but those undergoing operative delivery or instrument assisted vaginal deliveries tend to suffer greater morbidity. In this study, patients will be randomized to receive usual, guideline adherent, post-discharge care with or without a home nurse visit 1-2 days after nursery discharge. For each newborn and mother, information from the pregnancy, obstetrical record, and the nursery course will be collected. Data also will be recorded regarding continuity of care during the perinatal period, hospital readmissions, ED visits, compliance with and extent of outpatient care, satisfaction with and convenience of care, and costs of healthcare. Method of infant feeding, maternal confidence, maternal depression and anxiety, and satisfaction with care will also be assessed.

To accomplish the objectives of this project, we will focus on the following 3 specific aims:

SPECIFIC AIM 1. Establish that single home nursing visits improve healthcare delivery to and reduce adverse health outcomes for breastfeeding newborns.

This model of home visitation will be shown to reduce postnatal morbidities, improve compliance with post-discharge guidelines, and reduce disparities in health outcomes for those enrolled in a prospective trial based on data presented under Preliminary Studies conducted by the PI. A randomized, controlled trial will be conducted over a period of 36 months to demonstrate that infants that receive a single home visit have a reduced need for subsequent hospital-based or non-scheduled urgent care services. Secondary outcomes of importance will include compliance with follow-up guidelines and breastfeeding rates that also are expected to improve in those receiving a home visit.

SPECIFIC AIM 2. Establish that single home nursing visits improve healthcare delivery to and reduce adverse outcomes for mothers who are breastfeeding their newborns. Maternal readmission, emergency department utilization, and need for non-scheduled urgent care services will be reduced in the group of women receiving a single, postpartum home visit compared with standard care. Additionally, parenting sense of competence, satisfaction with postpartum healthcare, level of perceived social support, and the incidence of postpartum depression and anxiety will be improved among women randomized to receive a home nursing visit during the stressful and emotional period following childbirth compared with those randomized to not receive a home visit.

SPECIFIC AIM 3. Prospectively evaluate the cost-effectiveness of a single postnatal home nursing visit after maternity/nursery hospital discharge.

Data from the trial will be used to perform a stochastic cost-effectiveness analysis to demonstrate prospectively that a single home nursing visit is cost-effective based upon the reduction of the need for subsequent hospital or non-scheduled urgent care based services (inpatient, emergency department, and outpatient) for newborns and mothers in the first 14 postnatal/postpartum days. Again based on the previous retrospective study conducted by the PI, home visits are expected to be a cost-effective intervention. Other factors including maternal health outcomes, breastfeeding, and long-term health and social outcomes will be assessed in terms of their relationship with cost.

ELIGIBILITY:
Inclusion Criteria:

* Full term or late pre-term infant (> 34 0/7 weeks gestational age) discharged from the newborn nursery
* Feeding human milk (breast milk) during the maternity/newborn stay with intent to continue to breastfeed after discharge
* English speaking mother
* Singleton or twin infant

Exclusion Criteria:

* Premature infant < 34 weeks gestational age
* Exclusively formula fed infant during nursery stay
* Complicated maternity/nursery stay requiring > 2 night stay after a vaginal delivery or > 4 night stay after a cesarean section
* A nursery course with atypical complications (e.g. a work-up for ambiguous genitalia)
* Infant with hyperbilirubinemia requiring phototherapy during the nursery stay
* Any major maternal morbidities and/or pre-existing condition that would effect postpartum care such as cancer, multiple sclerosis, lupus, etc.
* Previous maternal participation in the NITTANY trial
* Residence outside of the coverage area for the Visiting Nurses Association (VNA) of Central Pennsylvania
* Family with no active telephone number (home or cellular)
* Infant being put up for adoption
* Non-English speaking mother
* Family requiring a home visit due to Social Work or other staff request/order
* Triplets or higher order gestation

Ages: 1 Day to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1154 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Use of unplanned maternal and child healthcare services (inpatient, Emergency Department (ED), urgent/acute care, primary care, and mental health) in the first 14 days after delivery | 3 years

SECONDARY OUTCOMES:
Adherence to continuity of care guidelines | 3 years
Postpartum anxiety | 3 years
Breastfeeding duration | 3 years
Maternal satisfaction with post-discharge healthcare | 3.5 years
Parenting sense of competence | 3.5 years
Cost of care | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State Milton S. Hershey Children's Hospital
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Hackman NM, Schaefer EW, Beiler JS, Rose CM, Paul IM. Breastfeeding outcome comparison by parity. Breastfeed Med. 2015 Apr;10(3):156-62. doi: 10.1089/bfm.2014.0119. Epub 2014 Dec 30. PMID 25549051
- [Derived] Paul IM, Downs DS, Schaefer EW, Beiler JS, Weisman CS. Postpartum anxiety and maternal-infant health outcomes. Pediatrics. 2013 Apr;131(4):e1218-24. doi: 10.1542/peds.2012-2147. Epub 2013 Mar 4. PMID 23460682
- [Derived] Bartok CJ, Schaefer EW, Beiler JS, Paul IM. Role of body mass index and gestational weight gain in breastfeeding outcomes. Breastfeed Med. 2012 Dec;7(6):448-56. doi: 10.1089/bfm.2011.0127. Epub 2012 Jun 25. PMID 23215909
- [Derived] Paul IM, Beiler JS, Schaefer EW, Hollenbeak CS, Alleman N, Sturgis SA, Yu SM, Camacho FT, Weisman CS. A randomized trial of single home nursing visits vs office-based care after nursery/maternity discharge: the Nurses for Infants Through Teaching and Assessment After the Nursery (NITTANY) Study. Arch Pediatr Adolesc Med. 2012 Mar;166(3):263-70. doi: 10.1001/archpediatrics.2011.198. Epub 2011 Nov 7. PMID 22064874
- See also: Penn State Milton S. Hershey Children's Hospital Pediatric Clinical Research Office — http://www.hmc.psu.edu/pedsclinicalresearch/index.htm